CLINICAL TRIAL: NCT03154710
Title: Relevance of a Web-mediated Follow up in Patients Having a Lymphoma With a High Risk of Relapse in Complete or Partial Response
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Negative interim analysis
Sponsor: Weprom (Other)
Collaborators: Sivan Innovation Ltd. (Industry); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ILC-1-2016; 2016-A01024-47 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-04

CONDITIONS: Lymphoma, T-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Hodgkin
Keywords: Web-mediated follow up; Lymphoma; Personalized medicine
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Lymphoma

STUDY DESIGN:
Intervention Model Description: Randomised, open, multicenter prospective trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-application follow up (Experimental): Patients will have a clinical and biological exam every 3 months and a web-mediated follow up. Patients will have to connect to the MOOVCARE application every 14 days to complete a questionnaire about their symptoms. Imaging will be performed in the event of an alert or clinical problem
  Interventions: Device: MOOVCARE
- Standard (No Intervention): Patients will have the usual follow up (Clinical and biological exam every 3 months and imaging every 6 months)

INTERVENTIONS:
Device: MOOVCARE — web-mediated follow up
  Arms: Web-application follow up

SUMMARY:
Lymphoma is the 6th cancer in terms of incidence in France where approximately 11,000 new cases are diagnosed each year. Most types of lymphomas occur at all ages with a predominance in elderly subjects.

With the continuous improvement of the diagnostic techniques and the treatments, the prognosis of lymphomas is constantly improving. However, 20-40% of patients relapse most often within 2 or 3 years after the end of treatment.

The current standard follow up includes a clinical examination and a biological check-up every 3 months for 2 years, then every 6 months up to 5 years and an imaging every 6 months. However, the interest of this systematic surveillance by imaging is controversial.

The use of new information and communication technologies, can improve the clinical follow-up of patients. To date, access to the Internet and portable technologies is sufficiently broad and democratized to envisage the use of this type of remote surveillance in the field of health. In particular to facilitate the dissemination of information between the patient and the physician. It is thus possible to imagine using this flow of information to generate alerts.

Strengthening the clinical follow-up in this indication, in which routine imaging has not demonstrated their interest, in particular by the implementation of remote monitoring completed by the patient, may present an advantage in terms of effectiveness and precocity of care. In this pathology, up to 40% of patients relapse early (within 2 to 3 years), in the vast majority of cases symptomatically (less than 2% asymptomatic relapse discovered by imaging). Finally the CT scan every 6-month , which generates radiation costs and exposures for a relatively low benefit, is performed in symptomatic patients since several weeks.

The aim of this study is to evaluate the interest of a web-mediated follow up using a score based on the dynamics and the association of clinical and biological signs to alert the physician of a possible recurrence of the patients treated for a lymphoma in complete or partial response.

DETAILED DESCRIPTION:
Lymphoma is the 6th cancer in terms of incidence in France where approximately 11,000 new cases are diagnosed each year. Most types of lymphomas occur at all ages with a predominance in elderly subjects.

With the continuous improvement of the diagnostic techniques and the treatments, the prognosis of lymphomas is constantly improving. However, 20-40% of patients relapse most often within 2 or 3 years after the end of treatment.

The current standard follow up includes a clinical examination and a biological check-up every 3 months for 2 years, then every 6 months up to 5 years and an imaging every 6 months. However, the interest of this systematic surveillance by imaging is controversial.

The use of new information and communication technologies, can improve the clinical follow-up of patients. To date, access to the Internet and portable technologies is sufficiently broad and democratized to envisage the use of this type of remote surveillance in the field of health. In particular to facilitate the dissemination of information between the patient and the physician. It is thus possible to imagine using this flow of information to generate alerts.

Strengthening the clinical follow-up in this indication, in which routine imaging has not demonstrated their interest, in particular by the implementation of remote monitoring completed by the patient, may present an advantage in terms of effectiveness and precocity of care. In this pathology, up to 40% of patients relapse early (within 2 to 3 years), in the vast majority of cases symptomatically (less than 2% asymptomatic relapse discovered by imaging). Finally the CT scan every 6-month , which generates radiation costs and exposures for a relatively low benefit, is performed in symptomatic patients since several weeks.

In addition, strengthened clinical follow-up may improve the early detection of relapses and also improve surveillance of all significant clinical complications commonly seen in patients with severe disease (sepsis, thromboembolism, late iatrogenics, etc.). If a benefit in survival is to be expected, it will most likely be due to the early detection of relapses and better control of recidivism through early treatment and management and the early implementation of appropriate supportive care, if only by the management of depressive symptoms, or the management of iatrogenic or other complications.

The aim of this study is to evaluate the interest of a web-mediated follow up using a score based on the dynamics and the association of clinical and biological signs to alert the physician of a possible recurrence of the patients treated for a lymphoma in complete or partial response.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with either:

   1. T-cell lymphoma in first complete or partial response
   2. Hodgkin lymphoma in 2nd complete or partial response including after autograft
   3. Large B-cell diffuse lymphoma in 2nd complete or partial response including after autograft
2. End-of-treatment imaging in the last 4 weeks
3. Age ≥ 18 years
4. PS ≤2 (WHO)
5. Patient with an initial symptoms score less than or equal to 5
6. Patient with internet access and mailbox
7. Patient affiliated to a social security scheme
8. Patient with written consent prior to any procedure specific to the study

Exclusion Criteria:

1. Patient whose lymphoma progressed at the end of the specific treatment (evaluation <3 months after the end of the previous treatment)
2. Symptomatic brain or meninges localisation
3. Presence or history of another cancer in the last 3 years, except skin cancers (other than melanoma), in situ cancers of the cervix or other cancers considered cured
4. Persons deprived of their liberty or under trusteeship
5. Dementia, mental impairment or psychiatric pathology that may compromise the informed consent of the patient and / or compliance with the protocol and follow-up of the study
6. Patients who can not follow the protocol for psychological, social, family or geographical reasons,
7. Pregnancy or breast-feeding
8. Patient participating in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katell LE DU, MD, Principal Investigator — Centre Jean Bernard - Le Mans
Locations (15):
- France (15):
  - CHBA Vannes, Vannes, Brittany Region
  - Institut Bergonié, Bordeaux, Gironde
  - Polyclinique du Parc, Caen, Normandy
  - Institut d'Hématologie de Basse Normandie, Caen, Normandy
  - Hôpital Privé du Confluent, Nantes, Pays de Loire
  - Centre Hospitalier Universitaire Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre Hospitalier Univeritaire, Dijon
  - CHU Grenoble, Grenoble
  - Centre Jean Bernard, Le Mans
  - Ch Mont de Marsan, Mont-de-Marsan
  - Centre d'Oncologie de Gentilly, Nancy
  - Hopital Saint Louis, Paris
  - Clinique Saint Anne, Strasbourg
  - Centre Hospitalier Universitaire, Tours

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Web-application Follow up | Standard
Started | 27 | 25
Completed | 20 | 20
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Web-application Follow up | Standard | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (14.4) | 64 (12.9) | 65 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 11 | 10 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Significant Complications Detected and Confirmed by a Medical Consultation Performed Outside the Standard Follow-up
Description: In the experimental group, identification of the absence of alert in case of complications and in the standard arm, identification of the absence of medical consultation (referring physician) in case of complications.
Time Frame: 6 months
Population: The results presented are those of the interim analysis planned for the first 40 patients included.
  A complete analysis will be done on all the patients (52) after incrementing all the data of the patients included in a second step.
Measure: Count of Participants; unit: Participants
Groups:
- Web-application Follow up: Patients will have a clinical and biological exam every 3 months and a web-mediated follow up. Patients will have to connect to the MOOVECARE application every 14 days to complete a questionnaire about their symptoms. Imaging will be performed in the event of an alert or clinical problem
  MOOVECARE: web-mediated follow up
Arm/Group | Web-application Follow up | Standard
Number analyzed (Participants) | 20 | 20
Participants | 9 | 2

2. Secondary Outcome: Complication Detection Time
Description: Time between the diagnosis of a complication and the nearest expected date of the subsequent follow-up programmed
Time Frame: 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Number of Complication Observed
Description: Collection of all complication presented by patients
Time Frame: 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Rate of Hospitalization for Vital Emergency
Description: Collection of serious adverse events
Time Frame: 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Sensibility of the Web-application
Description: Number of alerts triggered by the application in relation to the results of the systematic imaging or triggered by an alert
Time Frame: 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Compliance
Description: Number of assessement completed (usually 1 per 2 weeks) by patients
Time Frame: 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Performances Status (PS) at Relapse
Description: PS according to WHO
Time Frame: 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Quality of Life
Description: Completion of the quality of life questionnaire QLQ-C30 at baseline and after 3, 6, 9 and 12 months
Time Frame: up to 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Depression
Description: Completion of the "HUMEUR PhQ9" questionnaire at baseline and after 3, 6, 9 and 12 months
Time Frame: up to 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Satisfaction
Description: Completion of a questionnaire after 6 months
Time Frame: 6 months
Reporting Status: Not Posted

11. Secondary Outcome: Progression Free Survival
Description: Time between the diagnostic of partial or complete response and the diagnostic of relapse
Time Frame: 24 months
Reporting Status: Not Posted

12. Secondary Outcome: Overall Survival
Description: Time between the diagnostic of partial or complete response and the patient's death
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Web-application Follow-up: Patients will have a clinical and biological exam every 3 months and a web-mediated follow up. Patients will have to connect to the MOOVECARE application every 14 days to complete a questionnaire about their symptoms. Imaging will be performed in the event of an alert or clinical problem
  MOOVECARE: web-mediated follow up
Arm/Group | Web-application Follow-up | Standard
All-Cause Mortality (participants affected / at risk) | 2/27 | 1/25
Serious Adverse Events (participants affected / at risk) | 4/27 | 5/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Web-application Follow-up (N=27) | Standard (N=25)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
fever (General disorders) | 1 (1) | 0 (0)
falls (General disorders) | 0 (0) | 1 (1)
endometriel carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
influenza A (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03154710/Prot_SAP_000.pdf